CLINICAL TRIAL: NCT02857634
Title: Study of the Contribution of Confocal Microscopy Dual Band in the Management of Bladder Cancer
Brief Title: Confocal Microscopy Dual Band in the Management of Bladder Cancer
Acronym: HEXVISIO
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0035
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-08

CONDITIONS: Urinary Bladder Neoplasm
Keywords: Urinary Bladder cancer; diagnosis; Cellvizio Dual Band
MeSH Terms: conditions — Urinary Bladder Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Using PDD, urothelial lesions will be resected. The samples will be immediately investigated effect under confocal microscopy (Cellvizio dual band) in order to keep the fluoresceine effect. After confocal microscopy samples will be fixed in formalin and prepare for the pathologist that will confirm the diagnosis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bladder tumor resection
  Interventions: Device: Cellvizio dual band

INTERVENTIONS:
Device: Cellvizio dual band — Using fluorescence cytoscopy, lesions in the bladder will be resected. The samples will be immediately observed in order to keep the fluorescein effect under confocal microscopy (Cellvizio dual band). After confocal microscopy samples will be fixed in formalin and prepare for the pathologist that will confirm the diagnosis. The Cellvizio system can be used to observe a resected sample ex vivo, offering a cellular-level view of internal tissue. This technique allows the visualization of the microstructure of the tissue in real-time which may improve targeted sampling, provide earlier disease detection and help patient management. The Cellvizio system includes miniaturized optics, optical fiber bundles, high-speed scanning and advanced image processing components.

SUMMARY:
Bladder cancer is one of the most common cancer worldwide and the second most frequent urological cancer. The photodynamic diagnosis technique (PDD) currently used (Hexvix®) has improved tumor detection but with a high false positive rate. Indeed, the main limitation of the PDD is its lack of specificity, ranging from 35 to 66%. The association of this technique with new technologies such as the Cellvizio Dual Band featuring simultaneous dual wavelength illumination and detection, could improve the identification of tumoral lesions. The objective of this study is to demonstrate the efficacy of Cellvizio dual band technique for the diagnosis of tumors bladders.

ELIGIBILITY:
Inclusion Criteria:

* Patients having 18 years old or more
* Patients with a bladder carcinoma and with indication of tumor resection under Hexvix procedure.
* Patients giving consent to participate in the study

Exclusion Criteria:

-No consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients following a tumor resection of the bladder
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Determination of the nucleo-cytoplasmic ratio of cells | at inclusion
  In order to perform comparison between benign versus malignant cytology, significant differences between cytoplasmic areas and nuclear areas will be determine to stablish a value of nucleo-cytoplasmic ratio

SECONDARY OUTCOMES:
Number of neoplastic lesions identified by Cellvizio compared to number of lesions identified by pathology | through the study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Bonnal, MD, Principal Investigator — Service d'Urologie, Groupement des hôpitaux de l'Institut Catholique de Lille
Locations (1):
- Groupement des Hôpitaux de l'Institut Catholique de Lille, Lomme, Nord, France

IPD SHARING:
Plan to Share IPD: No